CLINICAL TRIAL: NCT04880486
Title: Effects of Weight Training With VR on Pulmonary Function, Exercise Capacity and Quality of Life in Out-Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Weight Training With VR in Out-Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ching-Hsia Hung, Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-108-038
Record Dates: First submitted 2021-04-14; First posted 2021-05-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: COPD; COPD Exacerbation; Pulmonary Rehabilitation; Weight Training; Virtual Reality; Muscle Strength; Pulmonary Function; Quality of Life; Readmission
Keywords: Acute exacerbation of chronic obstructive pulmonary disease; upper extremity weight training; virtual reality; exercise capacity; functional capacity; adherence rate of exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): usually care with extra health education on upper limb exercise
  Interventions: Other: Education
- Exercise group (Experimental): usually care with extra supervision upper limb exercise with VR
  Interventions: Other: Education; Other: Supervision upper limb weight training exercise with VR

INTERVENTIONS:
Other: Education — Usual pulmonary rehabilitation education and pharmacological therapies, and taught them some limbs exercise, using social application to contact and suggestion giving as supervision.
Other: Supervision upper limb weight training exercise with VR — Participant is supervised by physical therapist to conduct upper limb weight training exercise with VR.
  Arms: Exercise group

SUMMARY:
Using weight training with virtual reality can help after discharge patients of acute exacerbation of chronic obstructive pulmonary disease, which maintained their quality of life, and improved their exercise capacity, pulmonary function, readmission condition.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a type obstructive lung disease which had become the third leading cause of deaths worldwide. The main symptoms including dyspnea, coughing, sputum production and acute exacerbation of COPD (AECOPD). The physical activity level, muscle power, exercise tolerance and quality of life (QoL) would decline rapidly when an episode of AECOPD occurred, with the worsen of the pulmonary function and activities level, the patient would get weaker and mortality rate would increase. Pulmonary rehabilitation (PR) had become a common-used clinical programs which including (but not limit to) medication, education, psychological support, nutrition consultation and exercise interventions.

In PR programs, exercise had been specifically pointed out for its improvement of physical activity level and quality of life, however, the adherence rate of programs remains low due to lack of motivation and insufficient training effect. Previous interventions preferred aerobic exercise conducting in sitting position considering the long-term sedentary life style of patients. However, such an intervention demonstrated little effect on increasing muscle power of lower extremities, results in insufficient physical activity level and functional performance. Besides, the interventions are usually single and repeatedly limb movement exercise which fail to brings up interests and results in poor motivation of the patients. Literatures review has suggested the highly involvement of upper extremities which is strongly contributed to independently daily living. The implantation of virtual reality in PR program has gained attentions with its advantage of facilitate the motivation. Therefore, the study aims to conduct the muscle strength training including both upper and lower extremities with the combination of virtual reality (VR). Anticipated result expects to provide a research evidence of innovative pulmonary rehabilitation exercise intervention.

The study will recruited 30 participants who will be randomly divided into control and intervention group. Control group will receive routine pulmonary rehabilitation including medication and education, the research stuff will give a brief explanation of home exercise, and weekly telemedicine to follow the exercise intensity and provide conciliation. Intervention group will receive the routine medical care. Extra weight training program targeting on upper extremities with the VR headsets will be conducted with the accompany of the research stuff. 3 times a week for 8 weeks (as a 24-times interference totally) interventions with muscle strength, exercise capacity, pulmonary function and improvement of quality of life will be assess to investigate the training effects. Expected result including the progression of muscle strength, oxygen uptake level, as well as pulmonary performance. The implantation of VR will also improve the motivation to participant, which will further alleviate the symptoms and quality of life. It can also provide some research evidence for clinical therapist to conduct an individualized exercise prescription for COPD.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization due to acute exacerbation of chronic obstructive pulmonary disease in preceding 1-year history
* age was between 40 to 85 years old

Exclusion Criteria:

* having a pulmonary rehabilitation in the past 1 month
* comorbidities that don't suitable for pulmonary rehabilitation, such as, untreatable cardiovascular disease, sinus tachycardia (HR>120), hypertension at rest if not adequately controlled, resting systolic blood pressure < 90 mmHg, and exercise contraindication
* advanced cancer with fatigue syndrome
* can't follow the orders
* physical impairment
* psychological impairment

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | baseline
  using handhold dynamometer to test 5 motions for bilateral side for 3 times.
Muscle Strength | 4 weeks
  using handhold dynamometer to test 5 motions for bilateral side for 3 times.
Muscle Strength | 8 weeks
  using handhold dynamometer to test 5 motions for bilateral side for 3 times.
Muscle Strength | 12 weeks
  using handhold dynamometer to test 5 motions for bilateral side for 3 times.
Cardiopulmonary exercise function test | baseline
  using CPET to test for the maximal exercise performance of participant
Cardiopulmonary exercise function test | 4 weeks
  using CPET to test for the maximal exercise performance of participant
Cardiopulmonary exercise function test | 8 weeks
  using CPET to test for the maximal exercise performance of participant
Cardiopulmonary exercise function test | 12 weeks
  using CPET to test for the maximal exercise performance of participant

SECONDARY OUTCOMES:
Pulmonary function test | 4 times (baseline, 4 weeks, 8 weeks, 12 weeks)
  using spirometry to test for pulmonary function of participant FEV1/FVC in liter
Respiratory muscle force | 4 times (baseline, 4 weeks, 8 weeks, 12 weeks)
  using digital pressure Guage to test for inspiratory/expiratory muscle force of participant MIP/MEP in cmH2O
Quality of life questionnaire | 4 times (baseline, 4 weeks, 8 weeks, 12 weeks)
  using questionnaires of EuroQol-5 Dimension (EQ-5D) to test for the quality of life of participant EuroQol-5 Dimension (EQ-5D): 5 levels of health status description to measure quality of life, a higher level means a worsen outcome
Quality of life questionnaire | 4 times (baseline, 4 weeks, 8 weeks, 12 weeks)
  using modified Medical Research Council dyspnea scale (mMRC) questionnaire to test for the chronic obstructive pulmonary disease symptom of participants
  Modified Medical Research Council dyspnea scale (mMRC): score from 0-4 to measure the symptom severity of chronic obstructive pulmonary disease, a higher score means a worsen outcome;
Quality of life questionnaire | 4 times (baseline, 4 weeks, 8 weeks, 12 weeks)
  using chronic obstructive pulmonary disease assessment Test (CAT) questionnaire to test for the chronic obstructive pulmonary disease symptom of participants
  chronic obstructive pulmonary disease assessment Test (CAT): score from 0-40 to measure the symptom severity of chronic obstructive pulmonary disease, a higher score means a worsen outcome;
Quality of life questionnaire | 4 times (baseline, 4 weeks, 8 weeks, 12 weeks)
  using clinical chronic obstructive pulmonary disease questionnaire (CCQ) to test for the chronic obstructive pulmonary disease symptom of participants
  Clinical chronic obstructive pulmonary disease questionnaire (CCQ): score from 0-60 to measure the symptom severity of chronic obstructive pulmonary disease, a higher score means a worsen outcome;

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsia Hung, Ph.D, Study Chair — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided